CLINICAL TRIAL: NCT03108118
Title: Diaphragm Injury and Dysfunction During Mechanical Ventilation
Acronym: MYOTRAUMA
Status: Completed | Type: Observational
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Principal Investigator, Ewan Goligher, Intensivist, University Health Network, Toronto
Other Study IDs: 12-5582-B
Record Dates: First submitted 2017-04-04; First posted 2017-04-11 (Actual); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Respiratory Insufficiency; Diaphragm Injury; Mechanical Ventilation Complication
Keywords: Diaphragm dysfunction; Acute respiratory failure; Weaning
MeSH Terms: conditions — Respiratory Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Acute respiratory failure: We are enrolling patients who are intubated because of acute respiratory distress syndrome, pneumonia, septic shock, or severe acute brain injury (GCS ≤ 8 prior to intubation). This population is targeted for study because they are at relatively high risk of requiring prolonged mechanical ventilation.

SUMMARY:
This study is designed to evaluate the relationship between diaphragm activity during mechanical ventilation and the development of ventilator-induced diaphragm dysfunction (VIDD). Diaphragm structure, activity, and function are monitored longitudinally over the first 7 days of mechanical ventilation.

DETAILED DESCRIPTION:
Multiple factors are responsible for injury to the diaphragm during mechanical ventilation and critical illness. Suppression of respiratory drive and respiratory muscle activity can contribute to diaphragm dysfunction and increase the risk of prolonged mechanical ventilation.

The objective of this study is to determine whether diaphragm inactivity or injurious loading of hte diaphragm during mechanical ventilation leads to the development of diaphragm weakness. To address this question, we are monitoring the diaphragm longitudinally over the first week of mechanical ventilation.

Diaphragm activity is monitored by measurements of transdiaphragmatic pressure and diaphragm electrical activity. Diaphragm function is assessed by maximal transdiaphragmatic pressure generation and by measurements of diaphragm neuromuscular coupling. Diaphragm structure is assessed by daily ultrasound imaging.

Study measurments commence at enrolment (within 36 hours of intubation) and continue for the first 7 days of the study (or until extubation or death, if earlier).

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (>18) with acute respiratory failure receiving invasive mechanical ventilation for less than 36 hours diagnosed with any of the following conditions: acute severe brain injury; moderate or severe ARDS; septic shock; pneumonia

Exclusion Criteria:

* Predicted probability of remaining alive and on the ventilator on ICU day 7 is less than 50%
* Liberation from mechanical ventilation is expected/planned within 24 hours
* High cervical spine injury (C5 or higher)
* Receiving mechanical ventilation for neuromuscular disease
* Acute exacerbation of an obstructive lung disease
* Known esophageal varices or any other condition for which the attending physician deems an orogastric catheter to be unsafe
* Esophageal, gastric or duodenal surgical procedures within the last 6 months
* Received mechanical ventilation for > 48 hours in the preceding 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Critically ill patients who are receiving invasive mechanical ventilation for less than 36 hours.
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2013-06-25 (Actual); Primary Completion 2019-12 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
Diaphragm dysfunction | 7 days
  Diaphragm dysfunction will be defined as maximal transdiaphragmatic pressure < 30 cm H2O and/or maximal diaphragm thickening fraction < 20% at study completion

SECONDARY OUTCOMES:
Diaphragm thickness | 7 days
Diaphragm neuromuscular coupling | 7 days
Duration of inactivity (hours) | 7 days
Patient-ventilator asynchrony rate | 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Ewan C Goligher, MD, PhD, Principal Investigator — University Health Network, Toronto
Locations (2):
- Canada (2):
  - Mount Sinai Hospital, Toronto, Ontario
  - University Health Network, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jaber S, Petrof BJ, Jung B, Chanques G, Berthet JP, Rabuel C, Bouyabrine H, Courouble P, Koechlin-Ramonatxo C, Sebbane M, Similowski T, Scheuermann V, Mebazaa A, Capdevila X, Mornet D, Mercier J, Lacampagne A, Philips A, Matecki S. Rapidly progressive diaphragmatic weakness and injury during mechanical ventilation in humans. Am J Respir Crit Care Med. 2011 Feb 1;183(3):364-71. doi: 10.1164/rccm.201004-0670OC. Epub 2010 Sep 2. PMID 20813887
- [Background] Levine S, Nguyen T, Taylor N, Friscia ME, Budak MT, Rothenberg P, Zhu J, Sachdeva R, Sonnad S, Kaiser LR, Rubinstein NA, Powers SK, Shrager JB. Rapid disuse atrophy of diaphragm fibers in mechanically ventilated humans. N Engl J Med. 2008 Mar 27;358(13):1327-35. doi: 10.1056/NEJMoa070447. PMID 18367735
- [Result] Goligher EC, Fan E, Herridge MS, Murray A, Vorona S, Brace D, Rittayamai N, Lanys A, Tomlinson G, Singh JM, Bolz SS, Rubenfeld GD, Kavanagh BP, Brochard LJ, Ferguson ND. Evolution of Diaphragm Thickness during Mechanical Ventilation. Impact of Inspiratory Effort. Am J Respir Crit Care Med. 2015 Nov 1;192(9):1080-8. doi: 10.1164/rccm.201503-0620OC. PMID 26167730
- [Derived] Coiffard B, Dianti J, Telias I, Brochard LJ, Slutsky AS, Beck J, Sinderby C, Ferguson ND, Goligher EC. Dyssynchronous diaphragm contractions impair diaphragm function in mechanically ventilated patients. Crit Care. 2024 Apr 2;28(1):107. doi: 10.1186/s13054-024-04894-3. PMID 38566126